CLINICAL TRIAL: NCT04233671
Title: A Mindfulness and Peer Mentoring Program to Improve Adherence to Medication Assisted Treatment for Opioid Use Disorders- R61
Brief Title: Minds and Mentors Program (MiMP)- R61
Acronym: MiMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Alabama at Birmingham (Other); Tuscaloosa Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R61AT010802-01 (NIH)
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-05

CONDITIONS: Opioid-use Disorder; Medication Assisted Treatment; Substance Use Disorders
Keywords: Opioid Use Disorder; Mindfulness based therapy; cravings; relapse prevention; treatment retention; depression; stress; anxiety; cortisol; peer mentors
MeSH Terms: conditions — Opioid-Related Disorders; Substance-Related Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Interventional Study Model: Parallel Assignment
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness based relapse prevention and peer mentoring (Experimental): MiMP is a twelve week program, meeting once per week for 12 weeks for approximately two hours. Eight weeks are facilitated by a licensed counselor, and four weeks are facilitated by a peer mentor.
  Interventions: Behavioral: Mindfulness based relapse prevention and peer mentoring
- 12 Step Treatment Program Control (No Intervention): The control group will meet for 12 weeks for standard 12 Step Facilitation meetings.

INTERVENTIONS:
Behavioral: Mindfulness based relapse prevention and peer mentoring — Importantly, the treatment will utilize a group format. Group process can serve as a vital agent in breaking down client denial about drug abuse problems. Groups have also been shown to be suitable for treating problems commonly associated with substance abuse, including depression, isolation, and shame.
  Additionally, groups intrinsically have many rewarding benefits, including reducing isolation and enabling members to witness the recovery of others. The eight-week group therapy intervention is co-led by a licensed counselor and a peer mentor for eight weeks, then followed by group sessions led by peer mentors for an additional four weeks.
  Arms: Mindfulness based relapse prevention and peer mentoring

SUMMARY:
The proposed research effort will:

The purpose of this study is as follows:

1. Test the feasibility and acceptability of a twelve- week mindfulness based relapse prevention protocol in combination with peer mentoring in individuals with opioid use disorder who are on medication assisted treatment.
2. Determine whether participation in a combination of mindfulness based relapse prevention and peer mentoring in comparison with an attentional control group: a) improves adherence to MAT b) decreases relapse and cravings c) improves psychosocial outcomes such as depression, anxiety, stress and social support

DETAILED DESCRIPTION:
Although medication assisted therapy (MAT) for opioid use disorders (OUD) is safe and effective and is currently considered the gold standard for treating OUD, adherence to MAT regimens remains a challenge. The goal of the proposed study is to determine the effectiveness of a mindfulness-based intervention that also utilizes peer mentors in addition to professional substance abuse therapists (the Minds and Mentors program [MiMP]) in improving adherence to MAT for OUD and reducing relapse rates in a sample of individuals with OUD who are also on MAT versus a twelve-step facilitation (TSF) program. The MiMP is a twelve-week intervention that uses group therapy and meets once a week for about two hours for eight weeks with a professional substance abuse therapist; after the completion of eight therapist led sessions, participants will attend four weeks of group therapy sessions conducted by a peer mentor. The peer mentor will also attend the initial eight sessions with the therapist to establish rapport with participants. The control group will attend twelve weeks of a standard twelve-step facilitation program. This study will utilize an individually randomized group treatment design with ten participants in both the intervention and control groups. Data collection will occur at baseline, end of treatment, and at 3, 6, and 12- month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* At least 19 years old.
* Opioid Use disorder diagnosis based on Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-V) criteria in the past 30 days
* Currently receiving MAT for OUD (e.g. methadone, naloxone, naltrexone, and buprenorphine) from an established provider
* Are within maintenance phase of MAT (not actively detoxing)
* May meet criteria for a mood, anxiety, or other psychiatric disorder based on the DSM-V criteria. Participants on maintenance medications for a mood or anxiety disorder must be stabilized on medications for at least 2 weeks before therapy initiation
* Capable of reading and understanding English
* Able to provide written informed consent (i.e. no surrogate)
* Willing to commit to 8 group therapy sessions, baseline, and follow-up assessments for 12-months after the end of treatment (14- month total)

Exclusion Criteria:

* Significant cognitive impairment
* Women who are pregnant
* Actively suicidal or homicidal
* Active psychosis and/ or
* Unstable medical conditions that contraindicate proposed treatment

Subject exit criteria:

* Increases in alcohol or drug use leading to the need for a more intensive level of care (i.e., medical detoxification, inpatient)
* Newly developed active suicidal or homicidal ideation
* Inability to manage psychiatric symptoms within the inclusion/exclusion criteria of the study (i.e., need for the initiation of maintenance psychotropic medications; development of psychosis). If it is determined, based on clinical criteria, that a participant needs to be started on maintenance medications for anxiety, mood or psychotic symptoms during the study, they will be discontinued from the treatment trial
* Inability to return for therapy sessions due to incarceration or hospitalization lasting longer than four weeks.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mercy N Mumba, PhD, Principal Investigator — University of Alabama, Tuscaloosa
Locations (2):
- United States (2):
  - Pathway Healthcare, LLC, Birmingham, Alabama
  - Fritz Clinic, Homewood, Alabama

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We consented 43 participants total over the course of the study. However, participants were only considered enrolled in the study once they completed their baseline data collection and were ready to be randomized. Therefore, there were some participants who signed informed consent but did not follow through to complete baseline data collection. We had 21 participants who followed through and completed the baseline data collection. These were considered enrolled in the study.
Groups:
- Mindfulness Based Relapse Prevention and Peer Mentoring: MiMP is a twelve week program, meeting once per week for 12 weeks for approximately two hours. Eight weeks are facilitated by a licensed counselor, and four weeks are facilitated by a peer mentor.
  Mindfulness based relapse prevention and peer mentoring: Importantly, the treatment will utilize a group format. Group process can serve as a vital agent in breaking down client denial about drug abuse problems. Groups have also been shown to be suitable for treating problems commonly associated with substance abuse, including depression, isolation, and shame.
  Additionally, groups intrinsically have many rewarding benefits, including reducing isolation and enabling members to witness the recovery of others. The eight-week group therapy intervention is co-led by a licensed counselor and a peer mentor for eight weeks, then followed by group sessions led by peer mentors for an additional four weeks.
Period: Overall Study
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Started | 13 | 8
Completed | 8 | 4
Not Completed | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control | Total
Number analyzed (Participants) | 13 | 8 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.54 (11.93) | 40.38 (13.15) | 43.57 (12.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 9 | 4 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 12 | 6 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Male | 9 | 4 | 13
  Female | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Days Adherence to Medication Assisted Treatment
Description: The primary outcome variable is adherence to medication-assisted therapy (MAT), quantified as the number of days MAT was received as indicated during the last 4 weeks of the intervention period. We expect that this can be treated as a continuous variable in regression models.
Time Frame: Last 4 weeks of the intervention period
Population: comparing means for the number of days participants were adherent to MOUD at week 12 (end of intervention). These data are accurate. All participants in the mindfulness-based relapse prevention and peer mentoring arm reported taking medications for 28 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 8 | 4
days | 28 (0) | 23.25 (9.5)

2. Secondary Outcome: Feasibility of Mindfulness Based Relapse Prevention as Measured by Retention Rate
Description: Retention rate (the number of participants completing T4 divided by the number who were randomized for each treatment arm)
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 13 | 8
Participants | 8 | 4

3. Secondary Outcome: Acceptability and Adherence to Mindfulness Based Relapse Prevention as Measured by the Treatment Acceptability/Adherence (TAAS) Scale
Description: Scores on the TAAS are scored on a scale of 1-7. For ease of interpretation by our participants and for data entry purposes, we asked participants to rate the experience on a scale of 1-10. The composite sum score was used for each person. Therefore, scores ranged from 10 to 100. Higher numbers mean more treatment acceptability and adherence
Time Frame: 3 months - at the end of the 12 week intervention
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 8 | 4
score on a scale | 71 (5.6) | 78 (9.8)

4. Secondary Outcome: Satisfaction With the Intervention Program
Description: Satisfaction with the intervention program will be assessed with the 8-item Client Satisfaction Questionnaire (CSQ-8). The total score will be computed by adding the 8 items for a composite score. The range for composite scores is from 8-32. Higher numbers mean more satisfied the participant is with the program.
Time Frame: 3 months - at the end of the 12 week intervention
Population: data were present for this variable for 11 participants total. 1 participants did not provide data on this outcome variable.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 7 | 4
score on a scale | 28.9 (1.1) | 30.8 (7.4)

5. Secondary Outcome: Acceptability of the Intervention Programs
Description: Exit interviews were conducted with all participants to determine whether participants rated the intervention as acceptable. The number who rated each intervention as acceptable is reported.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 8 | 4
Participants | 8 | 4

6. Secondary Outcome: Relapse Rate (Number of Participants With Relapse) as Determined by Urine Drug Screen
Description: Relapse will be measured during the last 4 weeks of the intervention period as determined by Urine Drug Screen (UDS). Participants were only considered relapsed if they had opiates (outside prescribed MOUD) or any other illicit substance detected in the urine drug screen during the last four weeks of the 12-week intervention.
Time Frame: Last four weeks of the 12-week intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 8 | 4
Participants | 3 | 2

7. Secondary Outcome: Relapse Rate (Number of Participants With Relapse) as Measured Via Self-report
Description: Relapse will be measured via self-report utilizing the Timeline Follow-back (TLFB). The total number of participants who self-reported relapse during the last four weeks of the intervention period per treatment arm.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 8 | 4
Participants | 3 | 2

8. Secondary Outcome: Opioid Cravings as Measured by the Opioid Craving Scale
Description: Cravings as measured by the Opioid Craving Scale (OCS), a modification of the Cocaine Craving Scale will be utilized to assess opioid craving. The OCS consists of three items rated on a visual analog scale from 0-10. The total score is calculated by averaging the three items. Higher means scores represent more craving.
Time Frame: 6 months
Population: data were present for this variable for 10 participants total. 2 participants did not provide data on this outcome variable.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 7 | 3
score on a scale | 2.2 (0.9) | 3.9 (2.4)

9. Secondary Outcome: Social Support as Measured by the Community Assessment Inventory
Description: Social Support as measured by the Community Assessment Inventory (CAI) to assess perceived support. The original CAI contains 37 items covering support within four areas i.e., family living with and outside, friends, and communities, with items in each area summed to create the corresponding subscales. Lower scores indicate less support and higher scores indicate greater support. We will only evaluate community support for the current study (containing 13 items). Therefore, scores ranged from 13 to 52.
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 7 | 3
score on a scale | 35.7 (1.5) | 27.0 (4.9)

10. Secondary Outcome: Depression as Measured by the Patient Health Questionnaire
Description: Depression as measured by the Patient Health Questionnaire (PHQ-9), a 9-item self-report that measures depressive symptoms. The participant's score may range from 1- 27. The interpretation of the total score is as follows: 1-4, Minimal depression; 5-9, mild depression; 10-14, Moderate depression; 15-19, Moderately severe depression; 20-27, Severe depression. Higher numbers mean more depressive symptoms at 12 weeks post-end of intervention.
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 7 | 3
score on a scale | 8.6 (2.5) | 12.7 (6.4)

11. Secondary Outcome: Stress as Measured by the Perceived Stress Scale
Description: Stress as measured by the Perceived Stress Scale (PSS), a 10-item self-report of perceived stress. Scores may range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14 to 26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 7 | 3
score on a scale | 20.6 (1.5) | 25.7 (3.8)

12. Secondary Outcome: Anxiety as Measured by the Generalized Anxiety Disorder Scale
Description: Anxiety as measured by the Generalized Anxiety Disorder Scale (GAD-7), a 7-item self-report of anxiety. The score for the seven items ranges from 0 to 21. Scores of 5-9 represent mild anxiety, 10- 14 represent Moderate anxiety, and scores greater than 15 represent severe anxiety. Higher numbers indicate higher anxiety at 12 weeks post-end of intervention.
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
Number analyzed (Participants) | 7 | 3
score on a scale | 6.4 (1.8) | 12.7 (5.9)

13. Secondary Outcome: Feasibility of Mindfulness-based Relapse Prevention as Measured by Randomization Rate
Description: Randomization rate (the number of participants randomized divided by the number of participants who consented). Participants consented to hear about the study before screening for eligibility was conducted. This was based on how our protocol was written. Therefore, some of the people who consented did not end up meeting the eligibility criteria for the study, and therefore were not considered enrolled in the study. The difference between consented participants and the enrolled participants is due to the screen failures. Participants are also only considered randomized after they complete all baseline data collection, including providing biosamples. We have revised this protocol for the R33 phase to avoid the issue of screen failures after the consent process is completed.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Overall Number of Participants: This combines both treatment arms ie. mindfulness-based relapse prevention and peer mentoring and twelve-step facilitation.
Arm/Group | Overall Number of Participants
Number analyzed (Participants) | 43
Participants | 21

14. Secondary Outcome: Feasibility of Mindfulness-based Relapse Prevention as Measured by Enrollment Rate
Description: Enrollment rate (the number of participants who sign the informed consent form divided by the number who are approached). Participants consented to hear about the study before screening for eligibility was conducted. This was based on how our protocol was written. Therefore, some of the people who consented did not end up meeting the eligibility criteria for the study, and therefore were not considered enrolled in the study. The difference between consented participants and the enrolled participants is due to the screen failures. Participants are also only considered randomized after they complete all baseline data collection, including providing biosamples. We have revised this protocol for the R33 phase to avoid the issue of screen failures after the consent process is completed.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Number of Participants
Number analyzed (Participants) | 120
Participants | 43

15. Other Pre Specified Outcome: Baseline Cortisol Reactivity to Drug Cues
Description: Non-invasive salivary cortisol levels were assessed as a measure of stress reactivity to drug cues at baseline. A saliva sample was collected at baseline and again 20 minutes after watching a video depicting drug use. Saliva samples were assayed for cortisol levels. Cortisol reactivity for each participant was calculated using a difference score in which the baseline sample cortisol level was subtracted from the post-video sample cortisol level.
Time Frame: at baseline data collection
Measure: Mean (Standard Deviation); unit: microgram/dL
Groups:
- Mindfulness Based Relapse Prevention and Peer Support: MiMP is a twelve week program, meeting once per week for 12 weeks for approximately two hours. Eight weeks are facilitated by a licensed counselor, and four weeks are facilitated by a peer mentor.
  Mindfulness based relapse prevention and peer mentoring: Importantly, the treatment will utilize a group format. Group process can serve as a vital agent in breaking down client denial about drug abuse problems. Groups have also been shown to be suitable for treating problems commonly associated with substance abuse, including depression, isolation, and shame.
  Additionally, groups intrinsically have many rewarding benefits, including reducing isolation and enabling members to witness the recovery of others. The eight-week group therapy intervention is co-led by a licensed counselor and a peer mentor for eight weeks, then followed by group sessions led by peer mentors for an additional four weeks.
Arm/Group | Mindfulness Based Relapse Prevention and Peer Support | 12 Step Treatment Program Control
Number analyzed (Participants) | 8 | 4
microgram/dL | -.0837 (.132) | -.0045 (.063)

ADVERSE EVENTS:
Time Frame: 12-month period per participant.
Arm/Group | Mindfulness Based Relapse Prevention and Peer Mentoring | 12 Step Treatment Program Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-07-19): https://cdn.clinicaltrials.gov/large-docs/71/NCT04233671/Prot_SAP_ICF_000.pdf